CLINICAL TRIAL: NCT01370824
Title: Clinical Diagnosis Versus Histological Diagnosis by Punch Biopsy to Determine the Subtype of Basal Cell Carcinoma
Brief Title: Clinical Diagnosis of Basal Cell Carcinoma Subtype
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MEC 112041 (35344.068.11)
Record Dates: First submitted 2011-06-07; First posted 2011-06-10 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Basal Cell Carcinoma
Keywords: Diagnosis; Clinical; Punch biopsy; Surgical excision; Histology; Histopathology; Observed agreement; Diagnostic value; Accuracy; Interobserver variability; Intraobserver variability
MeSH Terms: conditions — Carcinoma, Basal Cell; Disease

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A punch biopsy and surgical excision of the BCC will be performed. Both biospecimens will be prepared with either frozen section histology, or paraffin embedded fixed tissue pathology.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Basal cell carcinoma: - Population: Eligible are patients (men and women) ≥18 years of age who visit the outpatient department of dermatology of the Maastricht University Medical Centre because of a clinically suspected BCC.
  - Inclusion criteria: All patients aged 18 years or older, otherwise healthy, with ≤ three primary (no previous treatment) clinically determined BCC.
  - Exclusion criteria: Patients using immunosuppressive drugs. Genetic skin cancer disorders. Earlier treatments at the same site. Age under 18 years. More than 3 clinical suspected BCCs. Not capable of informed consent.
  Interventions: Procedure: Punch biopsy; Procedure: Surgical excision

INTERVENTIONS:
Procedure: Punch biopsy — Punch biopsy is a 10 minutes treatment at the outpatient department of dermatology. Patient will lie down on a bed, the skin will be disinfected and local anaesthesia (lidocaine 1% with epinephrine) will be given, which is briefly painful. Then a PB of 3 mm is taken from the most suspected area. In the case of continuing bleeding the wound will be sutured. A properly taken biopsy will leave no or minimal scarring, but this is not relevant since a SE will be performed afterwards. In very rare cases post-biopsy bleeding or infection occurs.
Procedure: Surgical excision — Surgical excision takes place in 30 minutes. Patient will lie down on a bed, the skin will be disinfected and local anaesthesia will be given. sBCC and nBCC will be excised with a 3 mm margin, aBCC with a 5 mm margin. Most BCC can be surgically excised, but some have to be treated with Mohs micrographic surgery (MMS). MMS ensures total BCC removal, preserving as much surrounding skin with 100% margin control. All BCCs will be excised with a 2 mm margin and examined under the microscope. This will totally take 1.5-2.0 hours. If tumour is still present, another tissue layer with 2 mm margin will be excised. It usually takes removal of 1-3 tissue layers to complete MMS.
  After both treatments, wounds will be sutured and removed after 1-2 weeks, depending on the localisation. Within the first two weeks posttreatment, patients have to avoid physical heavy movements and keep the suture dry. Possible complications: scarring, continuous or subsequent bleeding, infection and dehiscent wounds.

SUMMARY:
Skin cancer is the most common cancer in Caucasians. Basal cell carcinoma (BCC) is the most frequent skin cancer with around 44.000 new tumours per year in the Netherlands, and its incidence is still rising. Prior to treatment, a punch biopsy (PB) is taken from the suspected lesion, in order to determine the subtype of BCC. There are three different histological subtypes of BCC, from least to most aggressive: superficial, nodular and aggressive. Based on the most aggressive subtype seen in the PB, a suitable surgical margin is chosen. Surgical excision (SE) is the treatment of first choice in all BCC subtypes according to the Dutch guidelines. Recent developments of non-invasive therapies for superficial BCC might be the first choice of treatment in the future. These non-invasive treatments (photodynamic therapy (PDT), Imiquimod and 5-fluorouracil (5-FU)) have better cosmetic results than SE and are therefore also used in the Maastricht University Medical Center. Drawback is a higher recurrence rate than SE. As nodular and aggressive subtypes grow deeper into the dermis, they have to be treated with SE with a 3 mm and 5 mm margin respectively. If BCC are located in the H-zone, the treatment will be Mohs micrographic surgery (MMS). Unfortunately, 30% of subtypes seen in the PB do not correspond with the subtype seen in the subsequent SE/MMS. The consequence is overtreatment and undertreatment. A potential better or equal way to determine the BCC subtype might be the clinical diagnosis. To our knowledge, there is no literature about the diagnostic value of the clinical diagnosis to determine the subtype of BCC seen in the SE/MMS specimen. We want to confirm the hypothesis that the clinical diagnosis is as good as, or even better than the histological diagnosis by PB to determine the BCC subtype in the subsequent SE/MMS. In this case, patients don't have to undergo an extra procedure, diagnostic route is shortened.

- Primary objective: to establish the observed agreement of clinical diagnosis compared to histological diagnosis by to determine the most aggressive subtype of BCC

- Secondary objectives: inter-observer and intra-observer variability of dermatologists and pathologists to determine subtype BCC.

DETAILED DESCRIPTION:
- Basal cell carcinoma throughout the world:

Skin cancer is the most common form of cancer, with basal cell carcinoma (BCC) being the most frequent form of all skin cancers, and the incidence is still rising without future signs of a plateau. Because there is no national registry for BCC in the Netherlands, incidence rates are derived from the only register centre in the southern part of our country. From a recent study we know that approximately 26.625 new patients with BCCs occurred in 2006 in the Netherlands. The average number of BCC per patient is 1.65, resulting in 44.000 new BCCs in that year. With an increase of approximately 10% per year the estimated incidence rate at 2011 will be around 70.800 in the Netherlands. Three important histopathologic subtypes of BCC can be distinguished, namely superficial, nodular and aggressive. In the past, nodular basal cell carcinoma (nBCC) was the most common histopathologic subtype, but superficial basal cell carcinoma (sBCC) and aggressive basal cell carcinoma (aBCC) are the subtypes with the fastest growing incidences. Nowadays, the distribution of histopathologic subtypes of BCC is 40.6% nodular, 30.7% superficial and 28.7% aggressive. The shift from nodular BCCs to other subtypes needs accurate detection of the correct subtype, as treatment per subtype is different. The sharp raising incidence of 10% annually makes BCC an even bigger health problem in the near future.

- Diagnosis of BCC:

BCC is diagnosed with a 3 mm punch biopsy (PB) of the suspected skin lesion. Based on the most aggressive histopathologic subtype seen in this biopsy, an appropriate treatment is chosen. Three subtypes are relevant for a suitable treatment choice: superficial, nodular and aggressive. The last one includes all BCCs with aggressive growth, such as infiltrative/morpheaform BCC, micronodular BCC, and BCC with squamous differentiation. Unfortunately, 31-33% of histopathologic subtypes seen on punch biopsies of primary and recurrent BCCs do not correspond with the subtype seen in the subsequent surgical excision (SE)/ Mohs micrographic surgery (MMS). The consequence is overtreatment and undertreatment.

- Guidelines on the treatment of basal cell carcinoma:

The national advisory board of Dutch dermatologists and plastic surgeons has published multidisciplinary guidelines on the treatment of BCCs in 2007. In these guidelines the different treatment options for all sort of BCCs are discussed and conclusions are drawn for each treatment option. Recommended treatments for all BCCs regardless of the histopathological subtype is SE. Both sBCC and nBCC have to be excised with 3 mm margin while aggressive subtypes need a 5 mm margin. BCCs in the H-zone will be excised with MMS. Photodynamic therapy (PDT), Imiquimod and 5-fluorouracil (5-FU) are also options for sBCC on low-risk sites because of better cosmetic results.Recent studies show overall estimated treatment success at 5-year follow-up of 65% for PDT and 78-80% for Imiquimod. These percentages are far lower than the 99% overall estimated treatment success of SE in sBCC. There is no literature on treatment effect of 5-FU at long term follow-up. Only two studies report 86-87% complete response rate to different 5-FU treatment regimens after 6-12 weeks.

- Treatment of basal cell carcinoma at the Maastricht University Medical Center (MUMC):

In the past, BCC has been a disease of the elderly patient but as a consequence of recreational sun exposure and tanning beds, more young patients develop a skin cancer as well. Therefore, cosmetic results play a more important role when choosing a suitable treatment. Therefore in today's dermatologic practice at the MUMC patients with a sBCC can be treated non-invasively with PDT, Imiquimod, 5-FU or with SE/MMS. These non-invasive treatments show good cosmetic results but higher recurrence rates than SE. Any non-responding or recurrent sBCC has to be retreated with SE/MMS.

- Undertreatment and overtreatment:

Preliminary data from our own study show that in case of a discrepancy between histopathologic BCC subtype in the PB and excision, 58% of patients are overtreated and 42% undertreated. Half of the overtreated patients will have a histological nBCC or aBCC on PB, but only superficial in the SE/MMS. This could be partly due to the fact that the most suspected part has already been biopsied and is not present in surgical excision anymore.

Overtreatment consists of unnecessary tissue loss because of too wide SE margins. In addition, large excisions might lead to more complications like scarring, infection, continued or subsequent bleeding and dehiscent wounds. Undertreated patients have to be re-treated again in case of positive resection margins with SE, resulting in extra stress for patients, time and health care costs.

- Clinical diagnosis:

Histological diagnosis of BCC subtype by PB might not be the perfect procedure because of the 30% mismatch with the subtype seen in the SE/MMS. A potential better way to determine the BCC subtype might be the clinical diagnosis. To our knowledge, there is no literature about the observed agreement of the clinical diagnosis to determine the most aggressive histological subtype of BCC. We want to confirm the hypothesis that the clinical diagnosis is as good as or even better than the histological diagnosis by PB to determine the most aggressive BCC subtype. Confirmation of this hypothesis will result in clinical diagnosis instead of punch biopsies, more patients receiving early and correct treatment, saving time and health care costs. The conclusions from the proposed study can serve as a basis for updating guidelines for the diagnosis of BCC.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years or older, otherwise healthy, with ≤ three primary (no previous treatment) clinically determined BCC will be recruited for this study.

Exclusion Criteria:

* Patients using immunosuppressive drugs. Genetic skin cancer disorders. Earlier treatments at the same site. Age under 18 years. More than 3 clinical suspected BCCs. Not capable of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible are patients (men and women) ≥18 years of age who visit the outpatient department of dermatology of the Maastricht University Medical Centre because of a clinically suspected BCC. The subtype will be determined by clinical diagnosis, histopathological examination of tissue derived from a PB and SE/MMS. Recruitment of the required number of patients (150 histological proven BCC, see below) should present no problems.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic value of clinical diagnosis | Within 24 hours after the patient presents at the outpatient department of dermatology
  The current proposal aims at establishing the observed agreement of the clinical diagnosis to and histological diagnosis to detect the most aggressive BCC subtype of the entire tumour.
Diagnostic value of punch biopsy | Histology within 2-3 weeks after the clinical diagnosis
  The current proposal aims at establishing the observed agreement of the clinical diagnosis to and histological diagnosis to detect the most aggressive BCC subtype of the entire tumour.
Diagnostic value of the surgical excision (SE)/ Mohs micrographic surgery (MMS) | Within 1 month after the punch biopsy
  The current proposal aims at establishing the observed agreement of the clinical diagnosis to and histological diagnosis to detect the most aggressive BCC subtype of the entire tumour.

SECONDARY OUTCOMES:
Interobserver and intraobserver variability | After clinical diagnosis, punch biopsy and surgical excision have been performed
  To assess the inter-observer and intra-observer variability of dermatologists and pathologists to determine subtype BCC.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole WJ Kelleners-Smeets, MD, PhD, Principal Investigator — Maastricht University Medical Center, Maastricht, the Netherlands; Ellen RM de Haas, MD, PhD, Principal Investigator — Erasmus Medical Centre, Rotterdam, the Netherlands
Locations (2):
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht, Limburg
  - Erasmus Medical Centre Rotterdam, Rotterdam